CLINICAL TRIAL: NCT00453622
Title: RISK Stratification Using a Combination of Cardiac Troponin T and Brain Natriuretic Peptide in Patients Receiving CRT-D
Acronym: RISK
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CRD303
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Resynchronization Therapy; Risk stratification; Prediction; Proteomics; Chemokine; cardiac enzymes; Brain Natriuretic Peptide
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy-Defibrillator — Implantation of a CRT-D device
  Other Names: CRT-D device

SUMMARY:
The purpose of the study is to identify if the combined use of cardiac troponin enzyme (cTnT) and brain natriuretic peptide (BNP) can predict Heart Failure (HF)improvement and all-cause mortality in patients implanted with cardiac pacemaker-defibrillation devices (CRT-D). Novel biochemical markers identifying patients with high risk cardiac mortality detected by plasma protein analysis will also be evaluated.

Hypothesis #1: The combined use of cTnT and BNP at just before implant will predict and risk stratify all cause mortality or HF hospitalization up to 12 months.

Hypothesis #2: The change in levels of said biomarkers at different points of follow-up can predict response to CRT through 12 months.

Hypothesis #3: The levels of a panel of novel inflammatory mediators, namely chemokines, will be correlated with improvement in 6-minute walk testing, quality of life, and left ventricular ejection fraction in CRT patients.

DETAILED DESCRIPTION:
Primary Endpoint

The primary endpoint is the occurrence of either death or first HF hospitalization. HF hospitalizations must satisfy both of the following criteria:

1. Admission to hospital for >24 hours with at least one of the following HF worsening symptoms:

   * Increased CHF class
   * Orthopnea
   * Paroxysmal nocturnal dyspnea
   * Edema
   * Dyspnea on exertion, or
   * Gastrointestinal (GI) symptoms attributable to HF
   * Placement on the Status I heart transplant list

   AND
2. One or more of the following intensive treatment(s) for HF within 24 hours of admission:

   * Intravenous (IV) diuresis
   * IV inotropic medications prescribed during the hospitalization, or
   * Increasing frequency of dialysis for patients with chronic renal failure

2.3 Secondary Endpoints

Secondary endpoints include:

* Cause of death
* Change in NYHA functional class
* Number of HF related hospitalizations
* Performance on a standard 6-minute hall walk test
* Quality of Life as measured by the Minnesota Living with Heart Failure (MLWHFQ) questionnaire
* Patient global clinical assessment
* Left ventricular ejection fraction (LVEF) measured by echocardiography
* LV volume measured by echocardiography
* LV lead placement position
* QRS duration at baseline and with CRT
* Number of AT/AF, VT/VF episodes
* Frequency of appropriate/inappropriate ICD therapy
* % Atrial and Ventricular Pacing
* Antiarrhythmic drug utilization
* Study related complications

2.3.1 Response to CRT

1. A positive response to CRT is defined by the following: Improvement in NYHA functional class by at least one grade
2. Improvement in echocardiographic LVEF & left ventricular end diastolic index (LVEDI)
3. Improvement in patient global clinical assessment
4. Improvement in 6-minute hall walk by 10%

ELIGIBILITY:
Inclusion Criteria:

* Referred for implantation of CRT-D according to currently accepted guidelines.
* 18 years or older
* Ability to independently comprehend and complete a QOL questionnaire
* Ability to provide informed consent for a study and be willing and able to comply with the prescribed follow-up
* Has stable conventional medications at least one month prior to enrollment

Exclusion Criteria:

* Inability to successfully implant an intravascular lead CRT-D device. (i.e. exclude epicardial leads)
* Myocardial infarction or unstable angina in the last 3 weeks
* Chronic atrial fibrillation (continuous AF lasting > 1 Month) within 1 year prior to enrollment or having undergone cardioversion for AF in the past month
* Status 1 classification for cardiac transplantation
* Currently participating in a clinical trial that includes an active treatment arm
* Life expectancy of less than 6 months.
* Recent (within 24 hours) administration of Nesiritide™

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart failure patients indicated for the CRT-D therapy
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2005-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
All Cause Death | 1 year follow up
First Heart Failure Hospitalization | 1 year follow up

SECONDARY OUTCOMES:
• Cause of death and ejection fraction | 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Aala Shalaby, MD, FACC, Principal Investigator — Veteran's Administration, Pittsburgh Healthcare System
Locations (1):
- Veterans' Adminstration Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Shalaby AA, Abraham WT, Fonarow GC, Bersohn MM, Gorcsan J 3rd, Lee LY, Halilovic J, Saba S, Maisel A, Singh JP, Sonel A, Kadish A. Association of BNP and Troponin Levels with Outcome among Cardiac Resynchronization Therapy Recipients. Pacing Clin Electrophysiol. 2015 May;38(5):581-90. doi: 10.1111/pace.12610. Epub 2015 Mar 30. PMID 25677851